CLINICAL TRIAL: NCT04596254
Title: Prospective Human Specimen Collection for Medical Research
Brief Title: Detection of Gut Metabolites in Mother's Milk Following Juice Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20.01.AMZ_BIO
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Healthy Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Juice Intake (Other)
  Interventions: Other: Pomegranate Juice

INTERVENTIONS:
Other: Pomegranate Juice — Collection of Mother's milk before and after juice consumption

SUMMARY:
The goal of the biological sample collection is to assess the presence of gut metabolites in human breast milk (BM) samples obtained prospectively from healthy lactating mothers and after consumption of fruit juice.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 yrs. female subjects with no lactation problems
* Healthy and term delivery
* Healthy dietary intake (vegetarian or omnivore)
* Agree to donate breast milk (not colostrum)
* First 6 months of lactation
* Subjects agree to consumer 8oz. of pomegranate juice for a week prior to 2nd collection

Exclusion Criteria:

* <20 yrs or >40 yrs. of age
* Subjects with lactation problems
* Preterm delivery
* Colostrum samples
* Lactation>6 months
* Subjects fail to drink juice for at least a week

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in levels of gut metabolites in breast milk following juice intake | 7 days
  Collection before and after juice intake

CONTACTS AND LOCATIONS:
Overall Officials: Anurag SIngh, MD, PhD, Study Director — Amazentis SA
Locations (1):
- Valleywise Health Biobank, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No